CLINICAL TRIAL: NCT05476445
Title: Comparison of the Effect of Cryotherapy Application and Low Level Laser Application on Post-Operative Pain in Primary Molar Teeth With Apical Periodontitis
Brief Title: Effect of Cryotherapy and LLLT on Postoperative Pain After Root Canal Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Muhammed Talha Çetin, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 28.04.2022/416
Record Dates: First submitted 2022-07-19; First posted 2022-07-27 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Root Canal Infection; Pain, Postoperative; Cryotherapy Effect; Laser; Pulpitis
Keywords: cryotherapy; LLLT; postoperative pain; pulpectomy; primary teeth
MeSH Terms: conditions — Pain, Postoperative; Pulpitis | interventions — Lasers; Cryotherapy

STUDY DESIGN:
Intervention Model Description: After the canal length was determined with the Apex locater, the canals were prepared using Ni-Ti endodontic rotary instrument files. Irrigation needles were kept 4-5 mm shorter than the working length, and irrigation of the channels was performed. A total of 5 ml of 1% NaOCl was washed for each canal, with 2 ml between each pecking movement of the files. The final washing of the channels was carried out using 5 ml of saline at room temperature.
  After the last wash, in the cryotherapy group, unlike the first two groups, each canal was washed with 5 ml of 2°C cold physiological saline for 5 minutes. After the canals were dried with the help of a paper cone, the canals were filled by injecting iodoform and calcium hydroxide-containing canals. Then the restoration was completed with compomer. Following the restoration in the LLLT group, the diode laser was activated in biostimulation mode for a total of 1 minute, 30 seconds in the buccal and lingual/palatal regions at the root apex.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients and the assessor don't know the study group names.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (Active Comparator): After the carious tissue was removed and the endodontic cavity was opened, isolation was provided with a rubber-dam. After the canal length was determined with the Apex locater, the canals were prepared using Ni-Ti endodontic rotary instrument files at the torque value recommended by the manufacturer in an endodontic motor. Irrigation needles were kept 4-5 mm shorter than the working length, and irrigation of the channels was performed. A total of 5 ml of 1% NaOCl was washed for each canal, with 2 ml between each pecking movement of the files. The final washing of the channels was carried out using 5 ml of saline at room temperature.After the canals were dried with the help of a paper cone, the canals were filled by injecting iodoform and calcium hydroxide-containing canals. Then the restoration was completed with compomer.
  Interventions: Procedure: Control
- Low level laser therapy (Experimental): After the carious tissue was removed and the endodontic cavity was opened, isolation was provided with a rubber-dam. After the canal length was determined with the Apex locater, the canals were prepared using Ni-Ti endodontic rotary instrument files at the torque value recommended by the manufacturer in an endodontic motor. A total of 5 ml of 1% NaOCl was washed for each canal, with 2 ml between each pecking movement of the files. The final washing of the channels was carried out using 5 ml of saline at room temperature.After the canals were dried with the help of a paper cone, the canals were filled by injecting iodoform and calcium hydroxide-containing canals. Then the restoration was completed with compomer. Following the restoration in the LLLT group, the diode laser was activated in biostimulation mode for a total of 1 minute, 30 seconds in the buccal and lingual/palatal regions at the root apex.
  Interventions: Procedure: Laser
- Cryotherapy (Experimental): After the carious tissue was removed and the endodontic cavity was opened, isolation was provided with a rubber-dam. After the canal length was determined with the Apex locater, the canals were prepared using Ni-Ti endodontic rotary instrument files at the torque value recommended by the manufacturer in an endodontic motor. Irrigation needles were kept 4-5 mm shorter than the working length, and irrigation of the channels was performed. A total of 5 ml of 1% NaOCl was washed for each canal, with 2 ml between each pecking movement of the files. The final washing of the channels was carried out using 5 ml of saline at room temperature.
  After the last wash, in the cryotherapy group, unlike the first two groups, each canal was washed with 5 ml of 2°C cold physiological saline for 5 minutes. After the canals were dried with the help of a paper cone, the canals were filled by injecting iodoform and calcium hydroxide-containing canals. Then the restoration was completed with compomer.
  Interventions: Procedure: Cryotherapy

INTERVENTIONS:
Procedure: Control — Root canal treatment
  Arms: Control
Procedure: Laser — Root canal treatment+Laser application
  Arms: Low level laser therapy
Procedure: Cryotherapy — Root canal treatment + Cryotherapy application
  Arms: Cryotherapy

SUMMARY:
The aim of this study is to evaluate the effect of low-level laser therapy (LLLT) and intracanal cryotherapy applications on postoperative pain in endodontic interventions of primary molar teeth with apical periodontitis. 75 patients were randomly assigned to the control, low-level laser and cryotherapy groups.Root canal treatments were performed in a single session. The pain intensity felt by the patients on the preoperative and postoperative 1st, 3rd, 5th and 7th days were recorded using the Wong Baker visual pain scale. Preoperative and postoperative 7th day percussion sensitivity was recorded using the VAS (visual analog scale) scale. The pain scores of the groups at different times after the procedure were compared. Statistical analysis of the data was performed at the 0.05 significance level.

DETAILED DESCRIPTION:
Patient Selection Criteria This study will be on primary molar teeth with acute pain at Atatürk University Faculty of Dentistry, Department of Pedodontics. While calculating the sample value, the effect value of Gundogdu et al.(2018) in terms of 1 day use in the evaluation was taken as 0.85, the standard deviation was 20, the α value was 0.05 and the β value was 95%, and the sample value was selected as 9 patients for each group. However, those who would be in good standing were in the unit 0.37 in the good group and in the 80% strong component, 0.05 significance elements were 75 samples for 3.

Treatment Protocol For treatment, 75 samples were first randomized with a web program (www.randemizer.org). According to this randomization, the incoming controls were separated from the leveled therapy (LLLT group) and intracanal cryotherapy (cryotherapy group) divisions (n=25).

The information about the data received for the study and the data related to the analysis are studied. Patients were treated by a single clinician.

The current pain intensity felt by the patients was determined using the Wong Baker visual pain assessment scale. In the evaluation of preoperative percussion sensitivity, a 10 cm VAS scale marked by the patient after the percussion test was used.

The teeth to be treated in each group were anesthetized using 1.8 ml of articain HCl (Ultracain DS; Pharma Vision San. ve Tic. A.Ş., Istanbul, Turkey) containing 1:100,000 epinephrine.After ensuring that anesthesia was provided, treatment was started.

After the carious tissue was removed and the endodontic cavity was opened, isolation was provided with a rubber-dam. #15 K files (Dentsply Maillefer, Ballaigues, Switzerland) were used to identify the root canals. After the pulp tissue in the canal was extracted with a tirnerf, the canals were washed with 2 ml of 1% NaOCl and dried using paper cones. The working length of the canals was determined using a #15 K file and electronic apex locator (Propex Pixi; Dentsply Maillefer, Ballaigues, Switzerland). After the working length has been determined, the canals are filled with Ni-Ti endodontic rotary instrument files (EndoArt Pedo Gold and EndoArt Expert Gold; İnci Dental Medical Malz. San. ve Tic. Ltd. Ş, Istanbul, Turkey) at the torque value recommended by the manufacturer, X Smart Plus ( Dentsply Maillefer, Ballaigues, Switzerland) was prepared using an endodontic motor.

In canals that could not be advanced passively up to the working length using a #20 K file, the canal length was measured with the #15 K file and 30.04 EndoArt Pedo Gold Ni-Ti endodontic rotary instrument file (İnci Dental Medical Malz. San. Ve Tic. Ltd. Şti, Istanbul, Turkey). ) has been prepared until. In the canals that cannot be progressed passively until the working length when the 25 numbered K file is used, the canal lengths were measured with the 20 numbered K file and 40.04 EndoArt Expert Gold Ni-Ti endodontic rotary instrument file (İnci Dental Medical Malz. San. Ve Tic. Ltd. Şti., Istanbul. ,Turkey) was prepared using. 30 gauge needles (Zhejlang Kangkang Medical-Devices Co.Ltd., Zhejlang, China) were preferred for use in canal irrigations. Irrigation needles were kept 4-5 mm shorter than the working length, and irrigation of the channels was performed. Irrigation was performed using 5 ml of 1% NaOCl in total for each canal, with 2 ml between each pecking movement of the files. Final irrigation of the canals was carried out using 5 ml of saline (0.9% Isotonic Sodium Chloride, Osel İlaç Sanayi ve Tic. A.Ş., Beykoz, Istanbul).

After the last irrigation, in the intracanal cryotherapy group, unlike the first two groups, each canal was washed with 5 ml of 2°C cold saline for 5 minutes. After the canals were dried with the help of a paper cone, the canals were filled by injecting iodoform and calcium hydroxide-containing canal paste (Viopex; Spident Co. Ltd, Incheon, Korea). After the paste residues on the cavity walls were cleaned with alcohol-impregnated cotton, resin modified glass ionomer cement (Ionoseal; Voco, GmbH, Cuxhaven, Germany) was placed on the pulp chamber floor and a LED light device (WoodPecker LED.B, Guilin Woodpecker Medical Instrument Co. Ltd, China) was used polymerized for 20 seconds. Dentin bonding agent (Futurabond U; Voco, GmbH, Cuxhaven, Germany) was applied to the cavity walls for 10 seconds, spread with light air for 5 seconds and then polymerized with light for 10 seconds. In the restoration of teeth, each layer of compomer (Figure 3.6., Twinky Star; Voco, GmbH, Cuxhaven, Germany) placed using the layering technique was light cured for 20 seconds. Following the occlusion control, polishing was done using green polishing rubber (OptraGloss, Ivoclar Vivadent Schaan, Liechtenstein) and the restoration process was completed.

After the restoration of the teeth is completed, unlike the other groups, in the LLLT group, the diode laser device (Diode Laser 3 Watt Expert03D810, China) biostimulation option was used in accordance with the user manual, at a wavelength of 980 nm, in continuous mode, 300 mW at the root apex level and 4 mm from the gingiva. It was activated for 30 seconds in the buccal region and 30 seconds in the lingual/palatal region. Before the DSLT application, protective glasses were used for patient and physician safety.

Painkillers (10 mg/kg paracetamol) were prescribed to all patients in case of very severe pain. Parents were asked to mark the patients' pain scores on the 1st, 3rd, 5th and 7th days according to the Wong Baker visual pain scale on the form given to the patients. The patients were called to a control appointment with the patient follow-up form they marked one week later. At the control appointment, the patients were asked whether they used painkillers after the procedure, and the presence of postoperative swelling, palpation and fistula tract was evaluated in their clinical examination and recorded in the form. In addition, the percussion sensitivity of the patients at the 7th day control appointment was determined using the VAS scale by performing the percussion test.

Statistical analysis After the data obtained in this study were recorded in Microsoft Excel program, statistical analyzes were performed in SPSS v26 program at p<0.05 significance level. Categorical variables were presented as numbers and percentages, and numerical variables as mean and standard deviation. Using the Kolmogrov Smirnov Test and the graphing method, it was evaluated whether the numerical variables were suitable for normal distribution or not. Chi-square test was used to compare categorical variables (gender, jaw, post-operative drug use and vitality) that did not show normal distribution. The numerical age variable with normal distribution was compared using one-way ANOVA. Kruskal Wallis test was used to evaluate more than two independent variables (pain difference between groups) that did not show normal distribution. More than two dependent variables (temporal variation of pain presence between groups) that did not show normal distribution were compared using Friedman analysis. The Willcoxon Sign test was used to evaluate two dependent variables (pain on the 1st, 3rd, 5th and 7th days within the groups) that did not show normal distribution.

In order to model the pain in the pain scores felt on the 1st and 7th days and the percussion sensitivity on the 7th day, the Binary Logistics regression analysis was performed with the Backward Conditional method using the relevant independent variables. The "no pain" group was taken as a reference in the analysis. The Hosmer-Lemeshow test result was evaluated in order to measure the effectiveness of the best model used to explain the dependent variable. The ratio of the independent variables in the model to explain the change in the dependent variable is shown by Cox and Snell and Nagelkerke statistics.

ELIGIBILITY:
Inclusion Criteria:

* The informed consent form is signed by the parent,
* The patient is between the ages of 6-9,
* The patient is cooperative (Frankl scale category 3 and 4),
* Having a history of spontaneous pain in primary molar teeth,
* Percussion sensitivity value before treatment is 5 or above 5 on the VAS pain scale,
* Presence of a primary molar tooth with acute or chronic infection in its pulp,
* When the crown pulp of primary molar teeth is removed, the bleeding in the root pulp does not stop or does not exist within 5 minutes,
* Primary molars that can be isolated with rubber-dam,

Exclusion Criteria:

* Patients with any systemic disease (including conditions requiring antibiotic prophylaxis) or psychiatric problems,
* Patients who used any analgesic, anti-inflammatory or antibiotic in the last 1 week in the last 24 hours before root canal treatment,
* Patients who are allergic to the materials used in the treatment,
* Primary molar teeth with excessive crown destruction that cannot be restored,
* Primary molar teeth with bone loss between roots exceeding 1/3,
* Having previously applied root canal treatment or amputation treatment in the relevant tooth,
* Presence of internal/external and physiological root resorption in the relevant tooth,
* Teeth with root fracture, ankylosis or mobility (Miller mobility classification 3 and 4),
* Teeth with excessive crown destruction that cannot be restored or a rubber-dam can be placed,

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2022-06-03 (Actual); Study Completion 2022-06-17 (Actual)

PRIMARY OUTCOMES:
Wong Baker wong baker faces pain rating scale | preoperative
  Patient's current pain. Scores between 0 to 5. Higher score means worse outcome.
Wong Baker wong baker faces pain rating scale | postoperative (1st day)
  Patient's current pain. Scores between 0 to 5. Higher score means worse outcome.
Wong Baker wong baker faces pain rating scale | postoperative (3rd day)
  Patient's current pain. Scores between 0 to 5. Higher score means worse outcome.
Wong Baker wong baker faces pain rating scale | postoperative (5th day)
  Patient's current pain. Scores between 0 to 5. Higher score means worse outcome.
Wong Baker wong baker faces pain rating scale | postoperative (7th day)
  Patient's current pain. Scores between 0 to 5. Higher score means worse outcome.
Visual Analog Scale (VAS) | preoperative
  Percussion pain of tooth. Scores between 0 to 10. Higher score means worse outcome.
Visual Analog Scale (VAS) | postoperative 7th day
  Percussion pain of tooth. Scores between 0 to 10. Higher score means worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Fatih Şengül, Phd, Study Director — Atatürk Uni. Faculty of Dentistry
Locations (1):
- Ataturk University Faculty of Dentistry, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gundogdu EC, Arslan H. Effects of Various Cryotherapy Applications on Postoperative Pain in Molar Teeth with Symptomatic Apical Periodontitis: A Preliminary Randomized Prospective Clinical Trial. J Endod. 2018 Mar;44(3):349-354. doi: 10.1016/j.joen.2017.11.002. Epub 2018 Feb 3. PMID 29398090
- [Background] Al-Nahlawi T, Hatab TA, Alrazak MA, Al-Abdullah A. Effect of Intracanal Cryotherapy and Negative Irrigation Technique on Postendodontic Pain. J Contemp Dent Pract. 2016 Dec 1;17(12):990-996. PMID 27965485
- [Background] Lopes LPB, Herkrath FJ, Vianna ECB, Gualberto Junior EC, Marques AAF, Sponchiado Junior EC. Effect of photobiomodulation therapy on postoperative pain after endodontic treatment: a randomized, controlled, clinical study. Clin Oral Investig. 2019 Jan;23(1):285-292. doi: 10.1007/s00784-018-2435-9. Epub 2018 Apr 16. PMID 29658070
- [Background] Arslan H, Doganay E, Karatas E, Unlu MA, Ahmed HMA. Effect of Low-level Laser Therapy on Postoperative Pain after Root Canal Retreatment: A Preliminary Placebo-controlled, Triple-blind, Randomized Clinical Trial. J Endod. 2017 Nov;43(11):1765-1769. doi: 10.1016/j.joen.2017.06.028. Epub 2017 Sep 28. PMID 28967495